CLINICAL TRIAL: NCT02338323
Title: Compare the Renal Protective Effects of Febuxostat and Benzbromarone in Chronic Kidney Disease Patients With GFR 20-50ml/Min
Brief Title: Compare the Renal Protective Effects of Febuxostat and Benzbromarone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ai Peng, Chief of department of Nephrology & Rheumatology, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FB2015
Record Dates: First submitted 2015-01-10; First posted 2015-01-14 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Chronic Kidney Disease; Hyperuricemia; Abnormal Renal Function
Keywords: Hyperuricemia; Renal Function; Chronic kidney disease; Febuxostat; Benzbromarone
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperuricemia | interventions — Febuxostat; Benzbromarone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Febuxostat (Experimental): take orally, 40mg per day, for 1 year
  Interventions: Drug: Febuxostat
- Benzbromarone (Experimental): take orally, 50mg per day, for 1 year
  Interventions: Drug: Benzbromarone

INTERVENTIONS:
Drug: Febuxostat — It acts as an inhibitor of xanthine oxidase, thus lowering urate concentrations in the body
  Other Names: Uloric; Adenuric
  Arms: Febuxostat
Drug: Benzbromarone — It is structurally related to the antiarrhythmic amiodarone, and it is a uricosuric agent and non-competitive inhibitor of xanthine oxidase
  Other Names: Desuric
  Arms: Benzbromarone

SUMMARY:
The purpose of this study is to determine whether febuxostat and benzbromarone could protect renal function, and which one could be better.

DETAILED DESCRIPTION:
Chronic kidney disease patients with hyperuricemia and glomerular filtration rate (GFR) 20-50 ml/min were treated by febuxostat or benzbromarone. Follow up the changes of serum uric acid, serum creatinine and GFR levels. Compare the effects on renal function of these two drugs.

ELIGIBILITY:
Inclusion Criteria:

Chronic kidney disease patients with glomerular filtration rate (GFR,20-50ml/min) who match one of the following criteria:

1. Gout
2. Hyperuricemia patients without gout but have cardiovascular risk and serum uric acid > 480umol/L
3. Hyperuricemia patients without gout but with serum uric acid > 540umol/L

Exclusion Criteria:

1. GFR<20ml/min or GFR >50ml/min
2. Liver dysfunction (Aspartate transaminase or/and alanine aminotransferase exceed 2 times of normal range)
3. Urinary tract obstruction
4. unstable angina, heart failure (stage III-IV, NYHA), new stroke, need diuretics for long-term treatment
5. Severe lung diseases or cancers
6. Pregnant woman or woman who prepare to be pregnant，nursing mothers
7. unable to sign informed consent form，or disagree with following-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Renal function | up to 12th months
  Blood test for serum uric acid and creatinine, according to equation to estimate glomerular filtration rate

SECONDARY OUTCOMES:
urine protein | 3rd months, 6th months, 9th months, 12th months
  urine test for microprotein markers and 24-hour urine protein quantitation
adverse drug reaction | 1st month, 2nd months, 3rd months, 6th months, 9th months, 12th months
  record all the adverse drug reactions

CONTACTS AND LOCATIONS:
Overall Officials: Ling Wang, MD, PhD, Study Chair — Department of Nephrology & Rheumatology, Shanghai Tenth People's Hospital
Locations (1):
- Department of Nephrology & Rheumatology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China